CLINICAL TRIAL: NCT03077724
Title: Fish Oil to Reduce Tobacco Use iN Expectant Mothers Study
Acronym: FORTUNE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Harvey Murff, Associate Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 161820
Record Dates: First submitted 2017-03-03; First posted 2017-03-13 (Actual); Results first posted 2019-01-09 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2018-12

CONDITIONS: Tobacco Use in Childbirth; Smoking Cessation; Pregnancy Related
Keywords: n-3 polyunsaturated fatty acids; tobacco use; pregnancy
MeSH Terms: conditions — Smoking Cessation; Tobacco Use | interventions — Fish Oils; Olive Oil

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, placebo controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, placebo control with medications dispensed by the Investigational Drug Service
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fish Oil (Experimental): 4.2 grams per day of n-3 long chain polyunsaturated fatty acids (LCPUFA)
  Interventions: Drug: Fish oil
- Placebos (Placebo Comparator): Olive oil supplements
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Fish oil — Fish oil supplementation
  Other Names: n-3 LCPUFAs
  Arms: Fish Oil
Drug: Placebos — Olive Oil capsules
  Other Names: Olive Oil
  Arms: Placebos

SUMMARY:
The purpose of this feasibility study is to obtain pilot data in preparation for an upcoming R01 submission. The goals of that submission will be to conduct a clinical trial of n-3 LCPUFAs for smoking cessation in pregnant women. For this proposal, the investigators will develop, test, and refine the recruitment strategy and collect data demonstrating the investigators ability to successfully recruit pregnant women who are actively smoking. The investigators will collect side effect, tolerability, and adherence data regarding the intervention. Finally, the investigators hope to gather preliminary effect size data to allow more formal estimates of sample size. The investigators hypothesize that pregnant smokers randomized to n-3 LCPUFA supplementation will have higher smoking cessation rates and less nicotine cravings compared to women allocated to placebo. The investigators intend to use this preliminary data to inform a future randomized, double-blind, placebo-controlled trial of n-3 LCPUFA supplementation for tobacco cessation.

DETAILED DESCRIPTION:
The goals of that submission will be to conduct a clinical trial of n-3 long-chain polyunsaturated fatty acids (LCPUFAs) for smoking cessation in pregnant women, who are at very high risk of continued smoking because pregnant generally cannot use any of the FDA-approved smoking cessation medications. Recently, two small scale, double-blind, randomized control trials have found that supplementation with n-3 LCPUFA reduces signs of nicotine dependence. While promising, these studies were not conducted in pregnancy, leaving an important gap in the scientific literature for this vulnerable group of smokers. For this proposal, the investigators will develop, test, and refine the recruitment strategy, and collect data demonstrating the ability to successfully recruit pregnant women who are actively smoking. The investigators will collect side effect, tolerability, and adherence data regarding the intervention. Finally, the investigators will gather preliminary effect size data on smoking behavior to allow more formal estimated of sample size for a larger, more definitive trial. The investigators hypothesize that pregnant smokers randomized to n-3 LCPUFA supplementation will smoke fewer cigarettes per day compared to women allocated to placebo. In secondary analyses the investigators will compare self-reported nicotine cravings and 7-day point-prevalence smoking abstinence (assessed at 30 days) between n-3 LCPUFA and placebo groups. The investigators intend to use this preliminary data to inform a future randomized, double-blind, placebo-controlled trial of n-3 LCPUFA supplementation for long-term tobacco cessation in pregnancy.

The specific aims are:

SA1: To successfully recruit and randomize 40 pregnant, current smokers into a clinical trial of n-3 LCPUFA supplementation.

SA2: To assess the tolerability of 4 gm/day n-3 LCPUFA supplementation in pregnant, current smokers over a 4-week period SA3: To determine the effect of 4 grams/day n-3 LCPUFA supplementation for 4-weeks on cigarettes smoked per day and self-reported nicotine cravings in pregnant smokers

Research Design and Methods This study is a randomized, double-blind, placebo controlled study of 4 grams/day n-3 LCPUFA supplementation versus placebo for 4-weeks. The study will recruit pregnant women in the second trimester who are currently smoking. The primary outcomes will include changes from baseline in cigarettes per day. The secondary outcome will be self-reported nicotine cravings, and point prevalence abstinence at 30 days. The investigators will also collect safety and tolerability data.

Eligible patients will be pregnant women who are currently smoking seen at Vanderbilt University Medical Center. The study is a single-site, randomized, double-blind, placebo-controlled, parallel arm trial design. The two arms included one treatment arm and one placebo arm. Treatment will be 4.2 grams/day of EPA + DHA. Placebo will be 5 grams of olive oil in capsule form. The intervention period will last 4-weeks. The study will randomize 40 participants into the two treatment arms. As this is a feasibility study, the investigators have not powered the study to account for drop-outs.

Participants will be identified through searching electronic searches, direct referral from the Tobacco Treatment Service, or self-referral from clinic fliers. Study physicians will conduct a medical chart review and participants who are potentially eligible will be invited for Clinic Visit 1 (baseline).

The study will include three clinic visits:

Clinic Visit 1: After eligibility is confirmed, consent will be obtained. A brief medical history will be obtained. Participants will complete five questionnaires. Subjects will complete the Fagerström Tolerance Questionnaire, the Minnesota Withdrawal Symptom Checklist, the Questionnaire of Smoking Urges-brief, the PHQ-4, and completes a detailed interview on tobacco use habits including recording cigarettes per day smoked. Questionnaires will be administered by study staff or CRC nurses directly into REDCap study databases. Blood, urine, and exhaled CO measurements will be collected. Participants will be dispensed a four-week supply of medication. Participants will be given a pill diary.

Clinic Visit 2: Participants will complete study questionnaires. Blood, urine, and exhaled CO measurements will be collected. Participants will report any adverse events.

Clinic Visit 3: Participants will complete study questionnaires. Blood, urine, and exhaled CO measurements will be collected. Participants will report any adverse events and return any unused medications.

Rationale for Dose:

As described above, two prior studies have been conducted in smokers to assess the effects of supplemental n-3 LCPUFAs on nicotine cravings. While both studies reported a statistically reduction in self-reported nicotine cravings in the intervention arms, a reduction in cigarettes smoked per day was only seen in the study of high-dose n-3 LCPUFA (> 4 grams/day) as opposed to low dose n-3 LCPUFA (1 gram/day). These studies would suggest a dose effect and as such the investigators are using a high-dose n-3 LCPUFA intervention for this pilot study.

Primary Outcome The primary outcomes will be reduction in total number of cigarettes per day from baseline to 4-weeks.

Secondary Outcomes The secondary outcome will be 1) reduction in the Fagerström Tolerance Questionnaire; and 2) point prevalence abstinence at 4 weeks biochemically confirmed by end-expired carbon monoxide.

Safety and Tolerability Outcomes Safety and tolerability outcomes will include: 1) reported AEs and 2) the rate of discontinuation of study medication due to side effects

Sample Size Justification and Statistical Analysis Plan Statistical analysis plan Descriptive statistics, including means, standard deviation, and ranges for continuous variables, as well as percent and frequencies for categorical variables, will be presented. Standard graphing and screening techniques will be used to detect outliers and to ensure data accuracy. For the primary analysis of post-intervention cigarettes per day, the investigators will perform a Wilcoxon (Mann Whitney) rank sum test evaluated at a 5% significance level. This data analysis plan will be carried out using statistical software SAS® (Cary, North Carolina) or statistical package R (R Development Core Team, 2008).

For the primary outcome the investigators will compare the change in total number of cigarettes smoked per day from baseline, 2-weeks, and 4-weeks. This outcome will be a continuous variable for this primary analysis. Secondary outcomes include the change in the Fagerström Tolerance Questionnaire, point prevalence abstinence at 4 weeks biochemically confirmed by end-expired carbon monoxide. The investigators will compare the change outcome at 4-weeks between arms using logistic regression using repeated measured ANOVA.

Sample size estimation and power analysis For the primary outcome, with the assumption of a baseline number of cigarettes per day of 11 with a SD of 5(11), the study should be able to detect a reduction by 41% in cigarettes per day in smokers allocated to the n-3 LCPUFA arm compared to placebo with 80% power.

The Fagerström Tolerance Questionnaire is on a 10-point Likert scale. Estimating a baseline score of 7.3 ± 1.6 the investigators have 80% power to detect a difference of 1 SD between the study arms.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 or ≤ 45 years of age
* Currently reporting daily cigarette use (≥ 1 CPD, no averages, must have daily use)
* Between 6 and 36 weeks gestation

Exclusion Criteria:

* Allergy to fish or seafood
* Currently using fish oil supplements and unwilling to stop prior to and during the trial
* Unstable psychiatric disease: Defined as requiring hospitalization or active medication changes (medication changes or up titration) within the preceding 3 months
* Unstable pregnancy-related medical problems (pre-eclampsia, premature labor, threatened abortion, oligohydramnios, placenta previa, hyperemesis gravidarum, HELLP syndrome, Intrauterine growth restriction, cholestasis of pregnancy, Rh negative disease, gestational hypertension, placenta accreta)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Eligibility requirements requires participant to be pregnant
Enrollment: 28 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2018-01-23 (Actual); Study Completion 2018-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harvey J Murff, MD, MPH, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
This is a pilot and feasibility trial. We are not planning to share IPD with other researchers

REFERENCES:
- [Background] Rabinovitz S. Effects of omega-3 fatty acids on tobacco craving in cigarette smokers: A double-blind, randomized, placebo-controlled pilot study. J Psychopharmacol. 2014 Aug;28(8):804-9. doi: 10.1177/0269881114536477. Epub 2014 Jun 4. PMID 24899596
- [Background] Zaparoli JX, Sugawara EK, de Souza AA, Tufik S, Galduroz JC. Omega-3 Levels and Nicotine Dependence: A Cross-Sectional Study and Clinical Trial. Eur Addict Res. 2016;22(3):153-62. doi: 10.1159/000439525. Epub 2015 Nov 17. PMID 26570994

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Olive oil supplements
  Placebos: Olive Oil capsules
Period: Overall Study
Arm/Group | Fish Oil | Placebo
Started | 14 | 14
Completed | 6 | 12
Not Completed | 8 | 2
Not completed — Lost to Follow-up | 5 | 1
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fish Oil | Placebo | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 32 [25 to 35] | 31 [28 to 34] | 31 [27 to 35]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 14 | 28
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 12 | 9 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 28
Marital Status [Count of Participants; unit: Participants]
  Married | 5 | 2 | 7
  Not Married | 6 | 11 | 17
  Separated/Widowed/Divorced | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Cigarettes Per Day From Baseline to 4-weeks
Description: Change in total number of cigarettes per day from baseline to 4-weeks
Time Frame: 4 weeks
Population: Participants with both baseline and 4-week complete data on cigarettes smoked per day
Measure: Median (Inter-Quartile Range); unit: Cigarettes smoked per day
Arm/Group | Fish Oil | Placebo
Number analyzed (Participants) | 6 | 12
Cigarettes smoked per day | -0.94 [-1.6 to 0.5] | 0 [-1.0 to 0]

2. Secondary Outcome: Change in Fagerström Scores From Baseline to 4-weeks
Description: Change in the Fagerström Test for Nicotine Dependency Score from baseline to 4-weeks. This scale is a validated instrument that measures nicotine dependency. The Fagerström Test for Nicotine Dependency is a 6-time survey. Each item is scores with a minimal score of 0 and a maximal score of 10. Higher scores indicate a higher level of nicotine dependency.
Time Frame: 4 weeks
Population: Change from baseline at 4-weeks in Fagerstrom scores
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Fish Oil | Placebo
Number analyzed (Participants) | 6 | 12
score on a scale | -1 [-2 to 0] | 0 [0 to 0]

3. Secondary Outcome: Point Prevalence Abstinence
Description: Point prevalence abstinence at 4 weeks biochemically confirmed by end-expired carbon monoxide
Time Frame: 4 weeks
Population: Subjects with complete baseline and 4-week measures
Measure: Count of Participants; unit: Participants
Arm/Group | Fish Oil | Placebo
Number analyzed (Participants) | 6 | 12
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: 1 month
Arm/Group | Fish Oil | Placebos
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 1/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fish Oil (N=14) | Placebos (N=14)
Hospitalization (Nervous system disorders) | 1 (1) | 0 (0) — Patient was on suboxone and noted after starting the study that she had lost her suboxone prescription. She presented to the emergency room and was admitted.

LIMITATIONS AND CAVEATS:
This was a feasibility study and the overall number of subjects was small. There was significant lost to follow up

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-26): https://cdn.clinicaltrials.gov/large-docs/24/NCT03077724/Prot_SAP_000.pdf